CLINICAL TRIAL: NCT04938674
Title: Application of Ultrasonic Guided Puncture in Blood Collection in Patients With Severe Trauma
Brief Title: Author-Wang Ping-- Research：Application of Ultrasonic Guided Puncture in Blood Collection in Patients With Severe Trauma
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0272
Record Dates: First submitted 2021-06-02; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2020-04

CONDITIONS: Severe Trauma
Keywords: ultrasound guidance; severe trauma; nursing care; blood specimen collection
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard process for blood collection using Ultrasonic Guided puncture
  Interventions: Device: ultrasonic guidance

INTERVENTIONS:
Device: ultrasonic guidance — Standard process for blood collection using Ultrasonic Guided puncture

SUMMARY:
This study aimed to investigate the application of ultrasound guided puncture technique in blood collection in patients with severe trauma. The methods of this study is 93 patients with severe trauma were selected from the emergency room of the Second Affiliated Hospital of Zhejiang University from April 2020 to September 2,2020 and from October 2020 to March 2021, comparing the differences between nursing treatment efficiency and doctor satisfaction.

DETAILED DESCRIPTION:
Standard process for blood collection using Ultrasonic Guided puncture.The control group used the traditional blood sample collection process, which was mainly based on personal clinical experience.

Statistical analysis using SPSS 25.0 statistical software. Observation index are time index of nursing treatment for patients with severe trauma: the time required for acquisition time, disposable puncture success rate, blood routine and blood type delivery time, rescue room stay time, etc and patient family and doctor satisfaction analysis: self-designed questionnaire, family satisfaction process, service time, service attitude, rescue technology, health education, including advice time, nursing quality, medical communication, teamwork, service attitude, evaluation levels: very satisfaction, satisfaction and dissatisfaction.

ELIGIBILITY:
Inclusion Criteria:

* ① airway obstruction, need tracheal intubation or intubation;② breathing stop, respiratory distress or significant slowing down;③ circulatory system shows various shock signs④GCS≤8;⑤ body table visible head, torso, chest open injury or yoke chest

Exclusion Criteria:

* All patients who stop the rescue room trauma evaluation and treatment midway through hospital transfer and automatic discharge

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with severe trauma received in the emergency room of the Second Affiliated Hospital of Zhejiang University Medical College from April 2020 to March 2021
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction analysis of the patient's family members | 1 year
  In contrast to the control group,patient family satisfaction survey includes medical time. The evaluation level is divided into 3 categories: very satisfied, satisfactory and unsatisfactory.
Time index of nursing treatment for patients with severe trauma | 1 year
  In contrast to the control group,time required for blood collection in patients with severe trauma
Satisfaction analysis of the doctors | 1 year
  In contrast to the control group,physician satisfaction survey includes executive advice time.The evaluation level is divided into 3 categories: very satisfied, satisfactory and unsatisfactory

CONTACTS AND LOCATIONS:
Overall Officials: Chen Ze Xin, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Zhejiang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No